CLINICAL TRIAL: NCT05236881
Title: Development of an mHealth Tool (ANíMATE) to Assess Self-management, Self-care and Adherence in People With Obesity
Acronym: ANíMATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-ANI-2020-10
Record Dates: First submitted 2022-01-24; First posted 2022-02-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-09

CONDITIONS: Obesity
Keywords: Obesity; mHealth; mobile application; self-management; self-care; adherence
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANíMATE mobile application (Experimental): Standard care protocol (3 face-to-face visits: basal, 2 and 4 months) + ANíMATE mobile application
  Interventions: Device: ANíMATE mobile application
- Standard care (No Intervention): Standard care protocol (3 face-to-face visits: basal, 2 and 4 months)

INTERVENTIONS:
Device: ANíMATE mobile application — mHealth tool ANíMATE (Adherence, Nutrition, PhysIcal Activity, Motivation, medicAtion, Technology and Empowerment) allows the recording of data related to diet and exercise and feedback on behavior through an intelligent data analysis system.
  Arms: ANíMATE mobile application

SUMMARY:
This trial main purpose is to develop and test an mHealth app aimed at improving self-management, self-care and adherence of people with obesity.

The study population are type I or II obese people, aged more than 18 years old, with or without comorbidities, who have a smartphone or tablet compatible with the app (Android version 9.0 or higher) and access to a scale for regular weight monitoring.

Control group will follow standard care protocol and patients in the intervention group will also be provided with the app. Follow-up will be done for 16 weeks. Both groups will attend 3 face-to-face visits (baseline, 2 and 4 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* People with BMI 30-39.9 kg/m2.
* Have a smartphone or tablet compatible with the app (Android version 9.0 or higher) and have sufficient capabilities to use it.
* Have access to a scale for regular weight monitoring.

Exclusion Criteria:

* Presence of serious major comorbidities: High blood pressure treated with > 3 drugs, diabetes mellitus treated with insulin, dyslipidemia treated with PCSK9 inhibitors, sleep apnea-hypopnea syndrome treated with CPAP, ischemic heart disease or stroke.
* Use of pharmacological treatment with influence on weight started in the 6 months prior to study entry.
* History of weight loss intervention (diet, exercise) in the 6 months prior to study entry.
* History of eating disorder.
* History of bariatric surgery.
* Use of any other app or treatment to lose weight in the 6 months prior to study entry.
* Pregnancy, short-term gestational desire or lactation.
* Any other disease or condition that may interfere with compliance with the protocol or completion of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
%TWL at 4 months | 4 months
  Percentage of total weight loss (%TWL) at 4 months

SECONDARY OUTCOMES:
%TWL at 2 months | 2 months
  Percentage of total weight loss (%TWL) at 2 months
%EWL at 2 and 4 months | 2 and 4 months
  Percentage of excess weight loss (%EWL) at 2 and 4 months
BMI change at 2 and 4 months | Baseline, 2 and 4 months
  Change in body mass index (BMI) (kg/m^2) from baseline to 2 and 4 months
Waist change at 2 and 4 months | Baseline, 2 and 4 months
  Change in waist circumference (cm) from baseline to 2 and 4 months
Blood pressure change at 2 and 4 months | Baseline, 2 and 4 months
  Change in systolic and diastolic blood pressure (mmhg) from baseline to 2 and 4 months
HbA1c change at 2 and 4 months | Baseline, 2 and 4 months
  Change in HbA1c percent from baseline to 2 and 4 months
Mediterranean diet adherence change at 4 months | Baseline and 4 months
  Change in mediterranean diet adherence questionnaire score (0*-14, *indicates worse questionnaire results) from baseline to 4 months
IPAQ change at 4 months | Baseline and 4 months
  Change in International Physical Activity Questionnaire (IPAQ) score (cathegory results: low/inactive*, moderate or high, *indicates worse questionnaire results) from baseline to 4 months
ACTA change at 4 months | Baseline and 4 months
  Change in attitudes towards change in eating disorders (ACTA) questionnaire score (0*-236, *indicates worse questionnaire results) from baseline to 4 months
Adherence to records | 2 and 4 months
  Percentage of records (weight, diet) at 2 and 4 months
Adherence to recommendations | 2 and 4 months
  Percentage of recommendations given by the medical team followed at next visit
Adherence to visits | 2 and 4 months
  Percentage of face-to-face visits attended
Adherence to the app | 2 months after the end of the study
  Percentage of patients who continue using the 2 months app after the end of the study
Quality of life change at 4 months | Baseline and 4 months
  Change in Short-Form Health Survey SF-36 questionnaire score (0*-100, *indicates worse questionnaire results) from baseline to 4 months
Satisfaction with the app | 4 months
  Satisfaction questionnaire in relation to the use of the app score (0*-20, *indicates worse questionnaire results) in the intervention group at the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain